CLINICAL TRIAL: NCT04358081
Title: A Multi-center, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety and Efficacy of Hydroxychloroquine Monotherapy and in Combination With Azithromycin in Patients With Moderate and Severe COVID-19 Disease
Brief Title: Hydroxychloroquine Monotherapy and in Combination With Azithromycin in Patients With Moderate and Severe COVID-19 Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJWT629A12301
Record Dates: First submitted 2020-04-08; First posted 2020-04-22 (Actual); Results first posted 2021-03-17 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Covid-19
Keywords: covid19; covid 19; covid-19; coronavirus; SARS-CoV; SARS-CoV-2; novel coronavirus; adult; JWT629; acute respiratory syndrome coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: hydroxychloroquine + aithromycin placebo (Experimental): Hydroxychloroquine 600mg o.d. as loading dose (Day 1) +followed by 200mg t.i.d was initiated within 8-12 hours of the loading dose (not to exceed 12 hours) Azithromycin (AZT) placebo o.d.
  Interventions: Drug: HCQ
- Arm 2: hydroxychloroquine + azithromycin (Experimental): Hydroxychloroquine 600 mg o.d. as a loading dose (Day 1) followed by 200 mg t.i.d. was initiated within 8-12 hours of the loading dose (not to exceed 12 hours) Azithromycin: 500 mg as a loading dose (Day 1) followed by 250 mg o.d. Day 2 - Day 5
  Interventions: Drug: HCQ+AZT
- Arm 3: hydroxychloroquine placebo + azithromycin placebo (Placebo Comparator): Hydroxychloroquine placebo o.d. (day 1) followed by hydroxychloroquine placebo t.i.d Azythromycin placebo o.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HCQ — Hydroxychloroquine Monotherapy
  Other Names: JWT629
  Arms: Arm 1: hydroxychloroquine + aithromycin placebo
Drug: HCQ+AZT — Hydroxychloroquine with azithromycin
  Other Names: JWT629 + AZT
  Arms: Arm 2: hydroxychloroquine + azithromycin
Drug: Placebo — Placebo
  Arms: Arm 3: hydroxychloroquine placebo + azithromycin placebo

SUMMARY:
Two recent studies have suggested that in patients with Covid19, treatment with hydroxychloroquine may shorten the duration of symptoms and improve viral clearance, an effect that appears most pronounced when combined with azithromycin. Hydroxychloroquine treatment may inhibit viral nucleic acid-mediated activation of various innate immune pathways, as well as blockade of lysosomal functions in cell types relevant for viral entry and antigen presentation.

The purpose of the study was to determine if oral hydroxychloroquine monotherapy, or in combination with azithromycin results in clinical benefit in patients hospitalized with COVID19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be obtained prior to participation in the study
2. Adult patient ≥ 18 years old
3. Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test from respiratory tract specimen (e.g nasopharyngeal swab)
4. Onset of signs and symptoms of COVID19 illness ≤ 7 days prior to randomization (including but not limited to fever, cough, myalgias, fatigue, abnormal chest imaging)
5. Currently hospitalized or requiring hospitalization due to COVID-19 disease

Exclusion Criteria:

1. Use of other investigational drugs or newly approved COVID-19 treatments within 5-half lives or 30 days of enrolment
2. History of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes
3. Participation in any other clinical trial of an experimental treatment for COVID-19
4. Expectation of concurrent treatment with any other agents or potential direct acting antiviral activity against SARS-Co V-2 during study drug dosing
5. Requires, in the judgement of the investigator, admission to the intensive care unit (ICU) or mechanical ventilatory support (invasive or non-invasive) prior to first dose of study drug (There might be a patient who cannot be admitted to the ICU, even if the patient's condition is severe enough, due to administrative reasons under the current circumstances. This case is also considered under admission to the ICU judged by the investigator)
6. Evidence of cytokine storm syndrome or multi-organ system failure
7. Confirmed co-infection with influenza
8. Creatinine clearance < 45 mL/min or requiring acute renal replacement therapy
9. History or current diagnosis of ECG abnormalities indicating significant risk of safety for participants participating in the study
10. Any other condition which in the opinion of the investigator, would put the safety of the participant at risk, impede compliance or hinder completion of the study
11. Pregnant or nursing (lactating) women
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they agree to use basic methods of contraception during dosing of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=859

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in 9 centers in the United States. A total of 20 participants were randomized, of whom 19 were treated.
Pre-assignment Details: One patient was mis-randomized and never received any treatment. This patient has creatine clearance level <45 mL/min or required acute renal replacement therapy and therefore was not eligible for inclusion in the study.
Groups:
- Arm 1: Hydroxychloroquine + Aithromycin Placebo: Hydroxychloroquine 600mg o.d. as loading dose (Day 1) +followed by 200mg t.i.d was initiated within 8-12 hours of the loading dose (not to exceed 12 hours) Azithromycin placebo o.d.
Period: Treatment Phase of Study
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo
Started | 7 | 7 | 5
Completed | 3 | 6 | 2
Not Completed | 4 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Period: Study Completion Phase
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo
Started | 7 | 7 | 5
Completed | 6 | 7 | 3
Not Completed | 1 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) was comprised of all participants to whom study treatment had been assigned by randomization excluding one mis-randomized participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo | Total
Number analyzed (Participants) | 7 | 7 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 5 | 16
  >=65 years | 0 | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (10.6) | 60.9 (12.5) | 55.2 (11.1) | 53.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 7
  Male | 4 | 6 | 2 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: FAS
  Participants
    White | 1 | 3 | 3 | 7
    Black or African American | 2 | 1 | 0 | 3
    Asian | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Unknown | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Clinical Response by Day 15
Description: Clinical response was defined as a) discharged alive; or b) No need for mechanical ventilation in any participants and no need for supplemental oxygen requirement (SpO2) in participants without pre-morbid O2 requirement.
Time Frame: 15 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo
Number analyzed (Participants) | 7 | 7 | 5
Participants | 7 | 7 | 4

2. Secondary Outcome: Number of Participants Who Achieved Viral Clearance
Description: Number and percentage of participants with negative or below LLOQ SARS-COV-2 based on polymerase chain reaction (PCR) test
Time Frame: 6 days and 10 Days
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Hydroxychloroquine + Aithromycin Placebo: Hydroxychloroquine 600mg o.d. as loading dose (Day 1) +followed by 200mg t.i.d was initiated within 8-12 hours of the loading dose (not to exceed 12 hours) Azithromycin (AZI) placebo o.d.
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo
Number analyzed (Participants) | 7 | 7 | 5
Participants
  by 6 days | 2 | 3 | 3
  by 10 days | 2 | 3 | 3

3. Secondary Outcome: Number of Participants Discharged or Ready for Discharge
Description: Number of participants who received hydrochloroquine plus azithromycin relative to placebo who were discharged from hospital
Time Frame: 15 days
Population: FAS
Measure: Number; unit: participants
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo
Number analyzed (Participants) | 7 | 7 | 5
participants | 7 | 7 | 4

4. Secondary Outcome: Time to Return to Pre-morbid Supplemental Oxygen Requirement in Participants Receiving Hydrochloroquine or Hydrochloroquine Plus Azithromycin Relative to Placebo
Description: Number of participants requiring supplemental oxygen at the time of randomization who returned to pre-morbid supplemental oxygen
Time Frame: 15 days
Population: FAS
Measure: Number; unit: participants
Arm/Group | Arm 1: Hydroxychloroquine + Aithromycin Placebo | Arm 2: Hydroxychloroquine + Azithromycin | Arm 3: Hydroxychloroquine Placebo + Azithromycin Placebo
Number analyzed (Participants) | 7 | 7 | 5
participants | 7 | 6 | 4

ADVERSE EVENTS:
Time Frame: at day 15
Description: Adverse Events (AEs) are any untoward sign or symptom that occured during the study treatment period of 15 days
Groups:
- Hydroxychloroquine + Aithromycin Placebo: HCQ
- Hydroxychloroquine + Azithromycin: HCQ + AZI
- Hydroxychloroquine Placebo + Azithromycin Placebo: HCG + AZI + Placebo
- Total: Total
Arm/Group | Hydroxychloroquine + Aithromycin Placebo | Hydroxychloroquine + Azithromycin | Hydroxychloroquine Placebo + Azithromycin Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 1/5 | 1/19
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 2/5 | 3/19
Other Adverse Events (participants affected / at risk) | 4/7 | 5/7 | 2/5 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxychloroquine + Aithromycin Placebo (N=7) | Hydroxychloroquine + Azithromycin (N=7) | Hydroxychloroquine Placebo + Azithromycin Placebo (N=5) | Total (N=19)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxychloroquine + Aithromycin Placebo (N=7) | Hydroxychloroquine + Azithromycin (N=7) | Hydroxychloroquine Placebo + Azithromycin Placebo (N=5) | Total (N=19)
Intracardiac mass (Cardiac disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 3
Pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 1
Neutrophil percentage increased (Investigations) | 0 | 1 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 2
Feeling of despair (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Only 20 participants of the initially planned 444 were randomized; and one of those was mis-randomized (so total of 19 participants). Due to this limited number of participants, study objectives could not be evaluated as planned. Results for select efficacy and for safety were summarized based in the information collected up to the eCRF database lock on 13-Aug-2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04358081/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT04358081/SAP_001.pdf